CLINICAL TRIAL: NCT05635734
Title: A Phase I/II Open Label Study to Assess Safety and Preliminary Evidence of a Therapeutic Effect of Azeliragon Combined With Conventional Concurrent Radiation and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: Azeliragon and Chemoradiotherapy in Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cantex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN 201; 2022-002801-36 (EudraCT Number)
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma
Keywords: Azeliragon; Newly diagnosed glioblastoma; Dose finding; Temozolomide; Radiotherapy
MeSH Terms: conditions — Glioblastoma | interventions — azeliragon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients will receive azeliragon for up to 2 years or as long as the patient and study investigator feel that a therapeutic benefit is possible.
  Patients will receive involved field radiation therapy and temozolomide consisting of fractionated focal irradiation in daily fractions of 2 Gy given 5 days/week for 6 weeks, for a total of 60 Gy, plus concomitant daily temozolomide (TMZ; 75 mg/m2/day, 7 days/week from the first to the last day of radiotherapy), followed by six cycles of adjuvant TMZ (150-200 mg/m2/day for 5 days during each of six 28-day cycles.
  Interventions: Drug: Azeliragon 5 mg; Drug: Azeliragon 10 mg; Drug: Azeliragon 20 mg

INTERVENTIONS:
Drug: Azeliragon 5 mg — Azeliragon 5 mg once a day (loading initial dose for 6 days of 10 mg daily). Patients will receive azeliragon for up to 2 years or as long as the patient and study investigator feel that a therapeutic benefit is possible.
  Patients will receive involved field radiation therapy and temozolomide consisting of fractionated focal irradiation in daily fractions of 2 Gy given 5 days/week for 6 weeks, for a total of 60 Gy, plus concomitant daily temozolomide (TMZ; 75 mg/m2/day, 7 days/week from the first to the last day of radiotherapy), followed by six cycles of adjuvant TMZ (150-200 mg/m2/day for 5 days during each of six 28-day cycles.
Drug: Azeliragon 10 mg — Azeliragon 10 mg once a day (loading initial dose for 6 days of 15 mg twice a day). Patients will receive azeliragon for up to 2 years or as long as the patient and study investigator feel that a therapeutic benefit is possible.
  Patients will receive involved field radiation therapy and temozolomide consisting of fractionated focal irradiation in daily fractions of 2 Gy given 5 days/week for 6 weeks, for a total of 60 Gy, plus concomitant daily temozolomide (TMZ; 75 mg/m2/day, 7 days/week from the first to the last day of radiotherapy), followed by six cycles of adjuvant TMZ (150-200 mg/m2/day for 5 days during each of six 28-day cycles.
Drug: Azeliragon 20 mg — Azeliragon 20 mg once a day (loading initial dose for 6 days of 30 mg twice a day). Patients will receive azeliragon for up to 2 years or as long as the patient and study investigator feel that a therapeutic benefit is possible.
  Patients will receive involved field radiation therapy and temozolomide consisting of fractionated focal irradiation in daily fractions of 2 Gy given 5 days/week for 6 weeks, for a total of 60 Gy, plus concomitant daily temozolomide (TMZ; 75 mg/m2/day, 7 days/week from the first to the last day of radiotherapy), followed by six cycles of adjuvant TMZ (150-200 mg/m2/day for 5 days during each of six 28-day cycles.

SUMMARY:
This is an open label study to determine the safety and preliminary evidence of a therapeutic effect of azeliragon in patients with newly diagnosed glioblastoma receiving concurrent radiation and temozolomide.

DETAILED DESCRIPTION:
Patients will receive involved field radiation therapy and temozolomide consisting of fractionated focal irradiation in daily fractions of 2 Gy given 5 days/week for 6 weeks, for a total of 60 Gy, plus concomitant daily temozolomide (TMZ; 75 mg/m2/day, 7 days/week from the first to the last day of radiotherapy), followed by six cycles of adjuvant TMZ (150-200 mg/m2/day for 5 days during each of six 28-day cycles.

Patients will receive azeliragon for up to 2 years or as long as the patient and study investigator feel that a therapeutic benefit is possible.

Patients will be accrued in groups of six starting with Dose Level 1. Escalation will continue as described in Table 2 until stopping rules are met or the highest defined dose level is reached. If Dose Level 1 is deemed intolerable, the trial will be closed to accrual.

The dose limiting toxicities (DLT) evaluation period will be defined as 28 days from initiation of dosing. The severity of adverse events will be graded according to CTCAE v 5.0. For the purpose of dose-finding, any listed AEs occurring during the DLT period, which are attributable (definite, probable, possible) to azeliragon will be classified as a DLT. In addition, the RP2/3D will take into account dose-reductions, treatment interruptions, discontinuation, and toxicities after the DLT period.

RP2/3D was defined as the dose with 6 patients treated at that dose level with ≤ 1 DLT observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically confirmed newly diagnosed glioblastoma (GBM, world health organization (WHO) grade IV). The histological diagnosis must have been made after biopsy or neurosurgical tumor resection.

   Note: Patients should be isocitrate dehydrogenase (IDH) wild type diagnosed locally
2. The local O-6-Methylguanine-DNA Methyltransferase (MGMT) report determination should be available and should be uploaded to the electronic case report form (eCRF).
3. Patient should have had a gross total or subtotal resection performed < 7 weeks prior to enrollment, documented at postoperative MRI. Patients who have had a biopsy only without resection are not eligible.
4. Patient deemed suitable by the treating physician to receive the standard radiotherapy regimen in combination with temozolomide.
5. Male or non-pregnant and non-lactating female and ≥ 18 to ≤ 70 years of age.
6. Patient may have received and continue to receive corticosteroids, but must be on a stable or decreasing dose for at least 14 days prior to first dose of study treatment.
7. Patient has not received prior chemotherapy or radiotherapy.
8. Patient has adequate biological parameters as demonstrated by the following blood counts at Screening (obtained ≤ 14 days prior to enrollment) and at Baseline-Day 0: Absolute neutrophil count (ANC) ≥ 1.0 × 109/L; Platelet count ≥ 75,000/mm3 (75 × 109/L); Hemoglobin (Hgb) ≥ 9 g/dL without transfusion or growth factor support
9. Patient has the following blood chemistry levels at Screening (obtained ≤ 14 days prior to enrollment) and at Baseline-Day 0:

   1. aspartate amino-transferase (AST)(SGOT), alanine transferase (ALT)(SGPT) ≤ 2.5 × upper limit of normal range (ULN). Total bilirubin ≤ 1.5 × ULN.
   2. Estimated creatinine clearance of > 60 mL/min (per Cockcroft -Gault formula)
10. Patients with a QTC of ≤ 480 msec
11. Patient has ECOG performance status of ≤ 2
12. Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form (ICF) prior to participation in any study-related activities.

Exclusion Criteria:

1. Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for > 5 years
2. Patients with a serious active infection (such as a wound infection requiring parenteral antibiotics) at the time of inclusion or other serious underlying medical conditions that would impair the ability of the patient to receive protocol treatment
3. Patients with any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.
4. Patients who have had treatment with any investigational cancer drug prior to the first dose of study treatment.
5. Patient has experienced an increase of ECOG to > 2 between Screening and the time of first dose with azeliragon.
6. Patients receiving CYP2C8 inhibitors
7. Patient is unwilling or unable to comply with study procedures, including, but not limited to self-administration of oral medication.
8. Patients with a gastrointestinal condition that could interfere with swallowing or absorption.
9. Females of childbearing potential who are sexually active or males with female partners of childbearing potential, where either the female or the male is unwilling to use a highly effective method of contraception during the trial and for 6 months after the last administration of azeliragon.
10. Patients with concurrent participation in another interventional clinical trial or use of another investigational agent within 14 days of starting azeliragon. Patients who are participating in non-interventional clinical trials (e.g., QOL, imaging, observational, follow-up studies, etc.) are eligible, regardless of the timing of participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2/3 dose | Throughout the DLT observation period, approximately 28 days per patient
  To assess the recommended phase 2/3 dose (RP2/3D) in mg/day of azeliragon in patients with newly diagnosed glioblastoma receiving concurrent radiation and temozolomide.
  Dose limiting toxicities were defined as listed AEs, dose-reductions, treatment interruptions, or discontinuation occurring during the DLT period (28 days), which are attributable (definite, probable, possible) to azeliragon will be classified as a DLT. 6 patients must be treated at that dose level with ≤ 1 DLT observed

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Throughout the study period, approximately 2 years per patient
  Percentage of patients experiencing an adverse event
Incidence of serious adverse events (SAEs) | Throughout the study period, approximately 2 years per patient
  Percentage of patients experiencing a serious adverse event
Disease control rate (DCR) | Throughout the study period, approximately 2 years per patient
  Percentage of patients who experience a complete response, partial response or stable disease according to Response Assessment in Neuro-Oncology (RANO) criteria as their best response throughout the study
Progression-free survival (PFS) | Throughout the study period, approximately 2 years per patient
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first
Overall survival (OS) | Throughout the study period, approximately 2 years per patient
  Defined as the duration of time from start of treatment to time of death
Patients with changes in the Eastern Cooperative Oncology Group (ECOG) performance status | Throughout the study period, approximately 2 years per patient
  Percentage of patients who experience a change in ECOG status through the study
S100A9 expression levels | Throughout the study period, approximately 2 years per patient in 3 occasions for each patient
  Expression levels of the S100A9 molecular biomarker in blood samples from patients. Samples will be taken at baseline, Week 10 and after progression

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sepúlveda, Study Chair — Hospital Universitario 12 de Octubre
Locations (4):
- Spain (4):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) anonymized could be shared upon request if the use is within the scope and protection level authorized by the patients by the signature of the informed consent

REFERENCES:
- [Derived] Comitre-Mariano B, Segura-Collar B, Vellila-Alonso G, Contreras R, Hernandez-Lain A, Valiente M, Sepulveda JM, Marcus SG, Garcia-Posadas G, Jimenez-Roldan L, Perez-Nunez A, Gargini R. S100A proteins show a spatial distribution of inflammation associated with the glioblastoma microenvironment architecture. Theranostics. 2025 Jan 1;15(2):726-744. doi: 10.7150/thno.100638. eCollection 2025. PMID 39744679